CLINICAL TRIAL: NCT04902625
Title: Use of Mysimba in Patients With Weight Regain After Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Nederlandse Obesitas Kliniek (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOK0023
Record Dates: First submitted 2021-05-18; First posted 2021-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-07

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Medication Persistence
Keywords: Bariatric Surgery; Anti-obesity Medication; Weight regain
MeSH Terms: conditions — Obesity, Morbid; Medication Adherence | interventions — Naltrexone-Bupropion combination; bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone-Bupropion combination (Active Comparator): The patients in this arm will receive 2 tablets of naltrexone-bupropion 8/90mg 2 times daily in combination with the Back On Track module.
  Interventions: Drug: Naltrexone-Bupropion Combination
- Control (No Intervention): The patients is this arm will only participate in the Back On Track module and will not receive any investigational or placebo product.

INTERVENTIONS:
Drug: Naltrexone-Bupropion Combination — Naltrexone-bupropion will be added to the BOT module in the interventional arm.
  Other Names: Mysimba; Contrave
  Arms: Naltrexone-Bupropion combination

SUMMARY:
Although bariatric surgery is currently the most effective treatment for morbid obesity, weight regain occurs in 16-37% of the patients (1). Weight regain is not regularly treated with antiobesity medications (AOMs).

Mysimba (Contrave in US) is a AOM, it is a combination of naltrexone hydrochloride extended release and bupropion hydrochloride extended release for the treatment of obesity, and is used with lifestyle modification. Bupropion is a mild reuptake inhibitor of dopamine and norepinephrine. Naltrexone, an opioid antagonist has minimum effect on weight loss on its own. Naltrexone is thought to block the inhibitory effects of opioid receptors activated by the β-endorphin released in the hypothalamus that stimulates feeding, thus allowing the inhibitory effects of α-melanocyte stimulating hormone to reduce food intake. In patients with obesity usage of Naltrexone/Bupropion (NB) results in up to 8.2% weight loss (2). There is some evidence that also in bariatric patients with weight regain NB leads to additional weight loss (3, 4).

At the Nederlandse Obesitas Kliniek (NOK) weight regain at follow-up is currently treated with the Back on Track (BOT) program. The BOT program is an extra intervention our clinic provides for the patients who have weight regain after surgery, this is part of our standard care program.

The primary objective is to study the effect of naltrexone/bupropion in combination with the BOT module on successful weight loss(>5% weight loss) after 22 weeks in patients with weight regain after bariatric surgery, compared to the regular BOT module.

DETAILED DESCRIPTION:
Throughout the years it has become clear that lifestyle intervention is the cornerstone for all types of bariatric treatment. Educating patients about behaviour, physical activity and intake strategies will help built a skills set, which patients can fall back on throughout their lives. Without additional lifestyle intervention a non-surgical, pharmacological or surgical treatment will be less effective. (5, 6) Besides lifestyle interventions, adjuvant pharmacological treatment has also proven to be effective in maintaining adequate weight loss. Pharmacological treatment is mostly performed in patients who are not eligible for bariatric surgery but do suffer from obesity and related comorbidities. Patients with a Body Mass Index(BMI) of ≥ 30kg/m2 or a BMI ≥ 27kg/m2 with an obesity-related comorbidity are advised to use pharmacological treatment. (7) In general the pharmacologic treatment affects appetite and therefore causes weight loss, provided that lifestyle interventions are added to the treatment.

For patients with a BMI of ≥ 40kg/m2 or a BMI ≥ 35kg/m2 with comorbid conditions bariatric surgery is advised. There is a variety of surgical treatment options, with Sleeve Gastrectomy (SG) and the Roux-en-Y gastric bypass (RYGB) being the most common. (8) An alteration of the gastro-intestinal tract is performed, which causes a change in gut hormones, bile acids and microbiota. These changes also have their effect on appetite and energy consumption causing an even higher weight reduction. (9) Although lifestyle interventions are the cornerstone of obesity treatment, bariatric surgery has proven to be a superior treatment. (9-11) Besides a positive effect on weight, bariatric surgery also has a positive effect on comorbidities, such as type 2 diabetes, hypertension, cancer incidence, cardiovascular events and cardiovascular deaths. (9, 10, 12-14) All in all we can state that bariatric surgery currently is the most effective treatment for patients suffering from morbid obesity.

Even though bariatric surgery is the most effective treatment, not all patients maintain their weight loss. As mentioned before weight regain occurs in 16-37% of the patients. (1) Currently these patients can be treated in our clinic with an extra module, the Back On Track (BOT) module. The BOT module consists of 4 extra sessions, 3 with the physiotherapist, psychologist or dietitian, and 1 with the medical doctor. During these sessions lifestyle modifications will once again be the main focus. A study performed with data from our own clinic shows an overall stabilisation of weight after this module. The regained weight will not be lost with the help of this module. Therefore other options should be explored.

One of the possibilities is the use of medication, in combination with lifestyle interventions (BOT module), to not only cause stabilisation of weight, but also weight loss at the end of our module.

Pharmacological therapy with other medication in post-bariatric patients is described to be a viable option. As described in the review performed by Sudlow et al, different medical options are being investigated. (15) At the moment most research has been focussing on pre-operative use of medication. In this review only four out of 20 studies described post-operative use of medication. Of these four only two studies researched the effect of naltrexone and bupropion combined in post-bariatric patients. Although these studies only have a small amount of participants (e.g. n=10), they do show a possible positive effect on weight loss. (3, 4, 15) Since there is a lack of research on the effect of pharmacotherapy as an addition to lifestyle interventions in post-bariatric patients, no clear guidelines can be created at the moment. (16)

Mysimba (Contrave in US) is Anti-Obesity Medication (AOM), it is a combination of naltrexone hydrochloride extended release and bupropion hydrochloride extended release. Naltrexone, mostly used for treatment of alcohol and opioid dependence, is thought to block the inhibitory effects of opioid receptors activated by the β-endorphin released in the hypothalamus that stimulates feeding, thus allowing the inhibitory effects of α-melanocyte stimulating hormone to reduce food intake. Bupropion is a mild reuptake inhibitor of dopamine and norepinephrine, which is used for treatment of depression and later for smoking cessation. On their own the effect on weight loss is minimal, when combined their effect on weight loss is synergistically positive. When combined with lifestyle interventions most successful results will be obtained.

In patients with obesity usage of Naltrexone/Bupropion (NB) has a stronger effect and results in up to 8.2% weight loss (2). A study performed by Apovian shows a significant difference in successful weight loss after 4 weeks, when comparing patients who use NB to patients with only lifestyle modifications. Their study had a follow-up period of 56 weeks with a extra measure timepoint at 28 weeks. All patients were measured and monitored every 4 weeks. The results at 4 weeks already showed a significant difference with the placebo group. (2) Furthermore, in a study conducted by Greenway et al after 16 weeks of follow up a significant difference in successful weight loss was observed. (17) So far not many studies have been conducted in post-bariatric patients. Even though the results thus far are scarce, they are promising. Two studies, both with a study population of 10, showed a positive result of around 5% more weight loss in post-bariatric patients. (3, 4)

In this study we will examine the effect of 2 tablets of Mysimba 8/90mg 2 times daily as addition to the Back On Track module for patients with weight regain after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI before surgery was ≥ 35,0 kg/m2
* Patient has undergone a primary banded/non-banded Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG)
* Gaining more than 5% weight after reaching plateau phase of lowest weight

Exclusion Criteria:

* Anatomical or surgical abnormalities for which revisional surgery is indicated.
* Use of the following medication Monoamino-oxidase inbibitors (MAO), selective serotonin reuptake inhibitor (SSRI), Tricyclic antidepressants (TCA), haloperidol, risperidone, opioids, antiarrhythmics, betablockers, antiviral medication (HIV)
* Pregnancy or breastfeeding
* Patients suffering from:

  * unregulated hypertension
  * a tumour in the central nervous system
  * severe liver failure
  * end stage kidney failure
* Patients suffering from or with a history of insults
* Patients with a history of:

  * bipolar disease
  * bulimia or anorexia nervosa
* Patients withdrawing from alcohol or benzodiazepines
* Patients who are not able to understand the informed consent form and patient information.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Effect naltrexone-bupropion in combination with the BOT module | 22 weeks
  The primary objective is to study the effect of naltrexone/bupropion in combination with the BOT module on successful weight loss (>5% weight loss) after 22 weeks compared with the regular BOT module alone, in patients with weight regain after bariatric surgery.

SECONDARY OUTCOMES:
Persistence | 22 weeks
  To describe the persistence of therapy of Mysimba after bariatric surgery. This will be described in amount of people completing the study with the full dosage or a lower dosage of Mysimba.
Tolerated dosage | 22 weeks
  To describe the maximal tolerated dosage
Adverse effects | 22 weeks
  To study adverse effects of the use of Mysimba
Weight loss | 12 months
  To monitor and compare weight loss more long term (up to 12 months) after the start of Mysimba in both study groups. Weight loss will be described in %Total weight loss.
Eating habits | 22 weeks
  To evaluate eating behaviour in patients with weight regain after bariatric surgery who used Mysimba compared to patients on the regular module according to the BODY-Q questionnaire
Medication absorption/exposure | 16 weeks
  a) To study bupropion and hydroxybupropion absorption/exposure by measuring steady-state serum levels in bariatric and compare these with steady-state serum levels in obese patients on Mysimba therapy who did not undergo bariatric surgery
Correlate serumlevels with effectiveness | 16 weeks
  b) to correlate bupropion and hydroxybupropion steady-state serum levels with effectiveness of Mysimba
Therapeutic range | 16 weeks
  c) to determine the therapeutic range of bupropion and hydroxybupropion plasma levels in bariatric and obese patients on Mysimba.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Greve, MD, PhD, professor, Principal Investigator — Nederlandse Obesitas Kliniek Zuid
Locations (1):
- Zuyderland Medical Center, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided